CLINICAL TRIAL: NCT05578651
Title: A Prospective, Single Center, Observational Study to Assess the Rapid Recovery After Cardiac Surgery Using SternaLock XP
Acronym: RACE XP
Status: Withdrawn | Type: Observational
Why Stopped: Zimmer Biomet has no current plans to market this product in EMEA.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 0821-02
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Rigid Plate Fixation; Median Sternotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SternaLock XP: Median sternotomy with rigid plate fixation (SternaLock XP) as the sole closure method
  Interventions: Device: SternaLock XP

INTERVENTIONS:
Device: SternaLock XP — Plating system with cable cerclage bands that is used in the stabilization and fixation of fractures of the anterior chest wall, including sternal fixation following sternotomy

SUMMARY:
The primary objective of this study is to evaluate the post-operative rapid recovery in patients treated with SternaLock XP for rigid sternal fixation with sternal precautions less restrictive than standard of care.

DETAILED DESCRIPTION:
The primary efficacy endpoint of evaluation is defined by the post-operative time back to prior work or life through patient diary.

The primary safety endpoint of evaluation is defined by the incidence rate of sternal complications (DSWI & SSWI) at 30 days post-op.

The secondary endpoints of evaluation up to 60-days post-operative are defined by:

* Quality of recovery after surgery (QoR-15)
* Days alive out of the hospital and at home (DAH)
* Disability-free survival (WHODAS 2.0.)
* Pain scores: Likert scale 1-10
* Opioid pain medication usage
* Spirometry: inspiratory vital capacity (IVC), as a measure of lung function recovery

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* ≥ 18 years of age, no upper limit
* Undergoing a full standard midline sternotomy as part of an elective or urgent cardiac surgical procedure [i.e., coronary artery bypass graft (CABG) and/ or valve replacement] and closed with the SternaLock XP Rigid Fixation System
* Willing to sign Informed Consent prior to the cardiac surgical procedure
* Willing and able to provide follow-up information up to 60-days post-operative

Exclusion Criteria:

Inclusion Criteria

* Male and female
* ≥ 18 years of age, no upper limit
* Undergoing a full standard midline sternotomy as part of an elective or urgent cardiac surgical procedure [i.e., coronary artery bypass graft (CABG) and/ or valve replacement] and closed with the SternaLock XP Rigid Fixation System
* Willing to sign Informed Consent prior to the cardiac surgical procedure
* Willing and able to provide follow-up information up to 60-days post-operative Exclusion Criteria

Pre-operative

* Emergent or salvage cardiac acuity, i.e., patients undergoing cardiopulmonary resuscitation en-route to the operating room or prior to induction of anesthesia
* Active or latent infection (with positive culture)
* Documented foreign body sensitivity, allergy, or intolerance to metals.
* Rapid bone absorption condition, metabolic bone disease, cancer, tumor, or tumor like condition of the bone, end-stage malignant disease, or other unexplained disease.
* Mental/ neurologic conditions rendering patients unwilling or incapable of following post-operative care instructions.
* Functional disability affecting gait, balance or mobility.

Operative

* Delayed sternal closure required for any reason (e.g., sent to ICU with open chest wound)
* Intra-operative conditions that, in the opinion of the operating surgeon, would preclude the use of rigid plate fixation.
* Insufficient quantity of sternal bone or limited blood supply as assessed by the operating surgeon using his or her professional judgment at the time of closure.
* Intraoperative death prior to device placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Received median sternotomy with rigid plate fixation after a cardiac procedure (e.g., valve replacement or repair, bypass grafting)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of sternal wound infection | 30 days
  Rate of deep sternal wound infection and superficial sternal wound infection

SECONDARY OUTCOMES:
Quality of recovery after surgery | 60 days
  QoR-15 instrument
Days alive and out of the hospital | 60 days
  Calculation of time
Disability-free survival | 60 days
  WHODAS 2.0 instrument
Pain score | 60 days
  Numerical Rating Pain Score
Opioid medication usage | 60 days
  Milligrams of morphine equivalency administered
Inspirometry vital capacity | 60 days
  Milliliters of spirometry capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Medical Center, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided